CLINICAL TRIAL: NCT06418464
Title: Efficacy and Safety of an Artificial-pancreas-like Learning-based Control in Type 1 Diabetes on Multiple Daily Injection Therapy: Protocol of a Multi-center, Non-inferiority, Randomized Controlled Trial (ELITE Study)
Brief Title: Efficacy and Safety of an Artificial-pancreas-like Learning-based Control in Type 1 Diabetes on Multiple Daily Injection Therapy
Acronym: ELITE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hebei Provincial People's Hospital (Unknown); Xingtai People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Liu, Associate Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023YFE0204100
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP-A Dosage Decision Support System (Experimental): The AP-A Dosage Decision Support System represents a new solution in diabetes care, offering customized insulin dosage recommendations to patients. This system is a product of integrating four pivotal modules: the individualized model learning module, the risk-sensitive control module, the Bayesian optimization module, and the safety constraint module. Together, they establish a robust framework that employs advanced computational methodologies to deliver precise and personalized insulin dosage guidance, significantly improving the effectiveness and safety of diabetes treatment plans. The actual injection dose in the intervention group was executed by the doctor after approval based on the recommendation of the AP-A Dosage Decision Support System.
  Interventions: Device: AP-A Dosage Decision Support System
- Physician decision-making (Active Comparator): The injection dose of the control group was determined by the doctor solely.
  Interventions: Device: AP-A Dosage Decision Support System

INTERVENTIONS:
Device: AP-A Dosage Decision Support System — The AP-A Dosage Decision Support System represents a new solution in diabetes care, offering customized insulin dosage recommendations to patients. This system is a product of integrating four pivotal modules: the individualized model learning module, the risk-sensitive control module, the Bayesian optimization module, and the safety constraint module. Together, they establish a robust framework that employs advanced computational methodologies to deliver precise and personalized insulin dosage guidance, significantly improving the effectiveness and safety of diabetes treatment plans. The actual injection dose in the intervention group was executed by the doctor after approval based on the recommendation of the AP-A Dosage Decision Support System.

SUMMARY:
This study is designed as a blinded, multi-center, non-inferiority randomized controlled clinical trial. It aims to enroll hospitalized T1D diabetes patients, ensuring an equal distribution with a 1:1 ratio between the intervention and control groups. The trial is set to take place across three locations in China: Peking University People's Hospital, Hebei Provincial People's Hospital, and Xingtai People's Hospital. Before participating, all subjects are required to provide their consent by signing a written informed consent form. Within the framework of the trial, the intervention group will receive insulin dosage recommendations from AP-A, subject to approval by a physician, whereas the control group will be treated with insulin dosages according to the current clinical guidelines established by their physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of an informed consent form.
2. Age between 18 and 70 years, with a T1D diagnosis of at least one year.
3. A confirmed diagnosis of T1D diabetes by at least two endocrinologists and fulfillment of at least one of the following conditions: a) Fasting C-peptide level less than 0.3 ng/mL. b) Fasting C-peptide level between 0.3 ng/mL and 0.6 ng/mL with at least one positive diabetic autoantibody.
4. Receiving intensified treatment regimen with multiple daily subcutaneous insulin injections upon screening and during the whole study period.

Exclusion Criteria:

1. Conditions such as diabetic ketoacidosis, diabetic ketosis, hyperglycemic hyperosmolar state, or other acute complications related to diabetes.
2. The presence of concurrent fever, severe infections, acute abdominal conditions, uncontrolled thyroid dysfunction, or the acute phase of any organ system disease.
3. A history within the last 3 months of serious cardiovascular issues including decompensated heart failure (NYHA Class III or IV), myocardial infarction, coronary artery bypass grafting, or coronary stent implantation, as well as uncontrolled severe arrhythmias or ischemic or hemorrhagic stroke.
4. Laboratory test abnormalities that exceed certain thresholds, such as alanine transaminase or aspartate transaminase levels greater than three times the upper limit of normal, total bilirubin levels more than twice the upper limit of normal, hemoglobin levels below 100 g/L, albumin levels below 30 g/L, or an estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73m².
5. Individuals who are required to fast or are unable to eat normally due to special circumstances.
6. Pregnant or breastfeeding women.
7. Individuals suffering from psychiatric illnesses or other cognitive impairments that may affect their ability to participate in the study.
8. Participants who are unable to wear a CGM due to severe allergies, skin diseases, or conditions at the sensor site such as lesions, scarring, redness, infection, or edema, which could interfere with the sensor's adhesion or the accuracy of glucose measurements in the interstitial fluid.
9. The systemic use of corticosteroids within the last month, with the exception of inhaled or topical steroids.
10. Any other condition or reason that the researcher deems to make the participant unsuitable for inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) | At the end of the treatment period
  The proportion of time that the glucose levels, as recorded by CGM during the treatment period, are within the range of 3.9mmol/L to 10.0mmol/L. This metric can be directly obtained by the algorithm system through closed-loop reading of CGM data.

SECONDARY OUTCOMES:
Time Below Range (TBR) | At the end of the treatment period
  The proportion of time that the glucose levels, as recorded by CGM during the treatment adjustment period, are below 3.9mmol/L.
Other Secondary Outcomes1 | At the end of the treatment period
  The proportion of glucose data stored by CGM during the treatment period that is in the range of 3.0-3.8mmol/L.
Other Secondary Outcomes2 | At the end of the treatment period
  The proportion of glucose data stored by CGM during the treatment adjustment period that is below 3.0mmol/L.
Other Secondary Outcomes3 | At the end of the treatment period
  The area under the curve (AUC) of glucose levels below 3.9mmol/L in the Ambulatory Glucose Profile (AGP) during the treatment adjustment period.
Other Secondary Outcomes4 | At the end of the treatment period
  The proportion of glucose data stored by CGM during the treatment adjustment period that is above 10.0mmol/L.
Other Secondary Outcomes5 | At the end of the treatment period
  The proportion of glucose data stored by CGM during the treatment adjustment period that is above 13.3mmol/L.
Other Secondary Outcomes6 | At the end of the treatment period
  The area under the curve (AUC) of glucose levels below 10.0mmol/L in the AGP during the treatment adjustment period.
Other Secondary Outcomes7 | At the end of the treatment period
  The mean of the glucose data stored by CGM during the treatment adjustment period (MEAN).
Other Secondary Outcomes8 | At the end of the treatment period
  The standard deviation of the glucose data stored by CGM during the treatment adjustment period (SD).
Other Secondary Outcomes9 | At the end of the treatment period
  The discrepancy between the physician-approved dosage and the AI-recommended dosage in the intervention group.
Other Secondary Outcomes10 | At the end of the treatment period
  The number of times the physician-approved dosage differs from the AI-recommended dosage in the intervention group.
Other Secondary Outcomes11 | At the end of the treatment period
  In the intervention group, the proportion of time that the glucose levels are within the range of 3.9mmol/L to 10.0mmol/L within 4 hours after insulin injection when there is a discrepancy between the physician-approved dosage and the algorithm-recommended dosage.

IPD SHARING:
Plan to Share IPD: Undecided